CLINICAL TRIAL: NCT02647346
Title: In-Home Assessment of a Smart Foot Mat for Prevention of Diabetic Foot Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Podimetrics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P-04
Record Dates: First submitted 2016-01-04; First posted 2016-01-06 (Estimated); Results first posted 2020-02-05 (Actual); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Foot Ulcer, Diabetic
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Participant cohort (Experimental): Participants with diabetes that each have a history of healed Diabetic Foot Ulcer (DFU) prior to enrollment.
  Interventions: Device: Daily use of podimetrics smart-foot mat

INTERVENTIONS:
Device: Daily use of podimetrics smart-foot mat

SUMMARY:
The purpose of this study is to investigate the accuracy of a Smart Foot Mat for signals associated with diabetic foot ulcers in high-risk patients.

ELIGIBILITY:
Inclusion Criteria:

* Male/Female, 18 years or older
* Diagnosis of type 1 or type 2 Diabetes Mellitus, controlled or uncontrolled
* Ankle Brachial Index (ABI) >0.5
* Patient with history of previous foot ulcer.

Exclusion Criteria:

* Active Charcot foot disease
* One or more plantar foot ulcers (UT Grade 1A-C, 2A-C & 3A-C)
* Active Infection/Gangrene
* Active malignancy
* Immunosuppressive disease
* History of alcohol or drug abuse
* Pregnant women (verbal confirmation or confirmation obtained within current medical records)
* Cognitive deficit
* 2+ or great lower extremity edema
* End stage renal disease
* History of major lower extremity amputation (below knee or above knee amputation)
* Other issue that, at the discretion of the investigator, renders the subject ineligible for participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2013-11; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Phoenix VA Health Care System, Phoenix, Arizona
  - University of Arizona, Tucson, Arizona
  - Center for Clinical Research Castro Valley, Castro Valley, California
  - Limb Preservation Platform, Fresno, California
  - VA Long Beach Health System, Long Beach, California
  - Miami VA Healthcare System, Miami, Florida
  - MetroWest Medical Center, Framingham, Massachusetts
  - Greenville Health System, Greenville, South Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Petersen BJ, Rothenberg GM, Lakhani PJ, Zhou M, Linders DR, Bloom JD, Wood KA, Armstrong DG. Ulcer metastasis? Anatomical locations of recurrence for patients in diabetic foot remission. J Foot Ankle Res. 2020 Jan 13;13:1. doi: 10.1186/s13047-020-0369-3. eCollection 2020. PMID 31956341
- [Derived] Frykberg RG, Gordon IL, Reyzelman AM, Cazzell SM, Fitzgerald RH, Rothenberg GM, Bloom JD, Petersen BJ, Linders DR, Nouvong A, Najafi B. Feasibility and Efficacy of a Smart Mat Technology to Predict Development of Diabetic Plantar Ulcers. Diabetes Care. 2017 Jul;40(7):973-980. doi: 10.2337/dc16-2294. Epub 2017 May 2. PMID 28465454

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Participant Cohort
Started | 132
Completed | 129
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Participant Cohort
Number analyzed (Participants) | 129
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 55
  >=65 years | 74
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 111
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Racial Origin: African American | 19
  Racial Origin: American Indian | 1
  Racial Origin: Asian | 2
  Racial Origin: Caucasian | 76
  Racial Origin: Hispanic/Latino | 26
  Racial Origin: Native American | 3
  Racial Origin: Unspecified | 2
Region of Enrollment [Number; unit: participants]
  United States | 129

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of Plantar Diabetic Foot Ulcer
Time Frame: Through study completion or subject withdrawal (34 weeks per-protocol)
Measure: Count of Participants; unit: Participants
Arm/Group | Participant Cohort
Number analyzed (Participants) | 129
Participants | 37

2. Secondary Outcome: Subject Adherence in Daily Use of the Study Device
Time Frame: Through study completion or subject withdrawal (34 weeks per-protocol)
Measure: Mean (Standard Deviation); unit: uses/week
Arm/Group | Participant Cohort
Number analyzed (Participants) | 129
uses/week | 5.5 (1.2)

3. Secondary Outcome: Device-related Trips/Falls
Time Frame: Through study completion or subject withdrawal (34 weeks per-protocol)
Measure: Number; unit: occurence
Arm/Group | Participant Cohort
Number analyzed (Participants) | 132
occurence | 0

4. Secondary Outcome: Device-related Injuries
Time Frame: Through study completion or subject withdrawal (34 weeks per-protocol)
Measure: Number; unit: occurence
Arm/Group | Participant Cohort
Number analyzed (Participants) | 132
occurence | 0

ADVERSE EVENTS:
Time Frame: 34 weeks
Description: Per the original definition of adverse event in the protocol, diabetic foot ulcer occurrence does not constitute as an adverse event.
Arm/Group | Participant Cohort
All-Cause Mortality (participants affected / at risk) | 3/132
Serious Adverse Events (participants affected / at risk) | 0/132
Other Adverse Events (participants affected / at risk) | 0/132

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No